CLINICAL TRIAL: NCT03882710
Title: Evaluation of Efficacy and Safety of Metoprolol XR in Patients Having Heart Failure With Normal Ejection Fraction: A Randomised, Double Blind,Placebo Controlled Trial
Brief Title: Metoprolol XR in Heart Failure With Normal Ejection Fraction
Acronym: HFNEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, SHotra, professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGI_Pharma_HFNEF 2010
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Diastolic Heart Failure
Keywords: heart failure, metoprolol, diastolic dysfunction
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoprolol XR capsule (Experimental)
  Interventions: Drug: Metoprolol XR
- placebo capsule (Placebo Comparator)
  Interventions: Drug: Metoprolol XR

INTERVENTIONS:
Drug: Metoprolol XR — Metoprolol XR capsule 25/50/100 mg once daily for 12 weeks
  Other Names: Metolar XL

SUMMARY:
In contrast to the treatment of HF with reduced EF, information to guide the pharmacological therapy of patients with HFNEF are lacking and there is no evidence based treatment for patients with HFNEF. Thus, present treatment strategies for HFNEF are largely based on assumptions regarding its pathophysiological mechanisms and on extrapolations from proven strategies used in systolic HF. Till now, no study enlightens the efficacy and safety of beta blockers in HFNEF in a randomised controlled manner although the role of beta blockers in HF with impaired systolic function has been sufficiently time tested leading to their therapeutic approval in that condition. Keeping in view the small reported benefit of beta blockers in HFNEF as mentioned above, there is a need to provide a conclusive proof of their role in this condition as well. Hence, investigators planned to test the efficacy and safety of metoprolol CR in patients with HFNEF in a randomised double blind placebo controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above of either sex
* Presence of New York Heart Association functional class II-IV of at least 4 weeks' duration
* LVEF ≥ 50% in a nondilated LV (LV end-diastolic volume < 97 ml/m2 measured by echocardiography)
* Echocardiographic evidence of LV diastolic dysfunction
* Willing to give written informed consent

Exclusion Criteria:

* Clinically unstable as defined by any change in diuretic dose in the month prior to enrolment.
* Significant valvular heart disease, pericardial disease, hypertrophic or restrictive cardiomyopathy
* Unstable angina or MI within the past 4 weeks.
* Alternative probable cause of the patient's symptoms (e.g.significant pulmonary disease);
* Any previous left ventricular ejection fraction below 40%
* Other systemic disease limiting life expectancy to less than 3 years
* Any contraindication to metoprolol use (heart rate less than 45 beats per minute, heart block greater than first-degree i.e. PR interval ≥ 0.24 second, systolic blood pressure <100 mm Hg, asthma)
* Conditions associated with alteration in serum levels of procollagen type I e.g. alcoholic liver disease, metabolic bone disease, hyperthyroidism
* Current participation (including prior 30 days) in any other therapeutic trial
* Any condition that, in the opinion of the investigator, may prevent the participant from adhering to the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing improvement of ≥ 1 in NYHA class | 12 weeks

SECONDARY OUTCOMES:
proportion of patients exhibiting any alteration in NYHA heart failure class from baseline | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Samir Malhotra, MD, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, UT-Chandigarh, India